CLINICAL TRIAL: NCT04684654
Title: A Double-Blind, Placebo-Controlled, Randomized, Single and Multiple Dose Study on the Safety, Pharmacokinetics, and Exploratory Pharmacodynamics of Subcutaneous and Intravenous BMS-986325 Administration in Healthy Participants and Participants With Primary Sjögren's Syndrome
Brief Title: BMS-986325 in Healthy Participants and Participants With Primary Sjögren's Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM039-004; 2019-003660-49 (EudraCT Number); U1111-1241-6583 (Other: WHO)
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy Participants; Primary Sjögren's Syndrome
Keywords: Primary Sjögren's Syndrome; Healthy participants; BMS-986325

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (SAD) (Experimental): Single Ascending Dose (SAD)
  Interventions: Biological: BMS-986325
- Part A (SAD) Placebo (Placebo Comparator)
  Interventions: Other: Placebo for BMS-986325
- Part B (MAD) (Experimental): Multiple Ascending Dose (MAD)
  Interventions: Biological: BMS-986325
- Part B (MAD) Placebo (Placebo Comparator)
  Interventions: Other: Placebo for BMS-986325
- Part C (pSS) (Experimental): Primary Sjögren's Syndrome (pSS)
  Interventions: Biological: BMS-986325
- Part C (pSS) Placebo (Placebo Comparator)
  Interventions: Other: Placebo for BMS-986325

INTERVENTIONS:
Biological: BMS-986325 — Specified dose on specified days
  Arms: Part A (SAD); Part B (MAD); Part C (pSS)
Other: Placebo for BMS-986325 — Specified dose on specified days
  Arms: Part A (SAD) Placebo; Part B (MAD) Placebo; Part C (pSS) Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, and drug effects of BMS-986325 in healthy participants and participants with primary Sjögren's syndrome. The results will guide the future clinical development with BMS-986325.

ELIGIBILITY:
Inclusion Criteria:

Healthy Participants (Part A and Part B)

* Healthy male and female participants as determined by no clinically significant deviation from normal in medical history, physical examination (PE), electrocardiograms (ECGs), and clinical laboratory determinations
* Males and Females, ages 18, or local age of majority, to 50 years, inclusive at screening
* Body mass index (BMI):18.0 to 30.0 kg/m2, weight: ≥ 50 kg at screening
* Must be fully vaccinated against SARS-CoV-2

Participants with Sjögren's Syndrome (Part C)

* Sjögren's syndrome in the absence of another immune-mediated disease or rheumatologic condition based on the 2016 American College of Rheumatology-European League Against Rheumatism (EULAR) Classification Criteria for primary Sjögren's syndrome (pSS). Historical diagnosis as pSS documented in medical records, using the 2016 ACR/EULAR criteria, is also acceptable
* Seropositive for anti-Sjögren's syndrome antigen A antibody (anti-SSA). Previous anti-SSA are also acceptable, and results should be documented in the Case Report Form (CRF) as past medical history
* Males and females, ages 18, or local age of majority, to 75 years, inclusive at screening
* Body mass index (BMI): 18.0 to 35.0 kg/m2; weight ≥ 50 kg at screening
* Must be fully vaccinated against SARS-CoV-2 according to local regulations

Exclusion Criteria:

Healthy Participants (Part A and Part B) - Any significant acute or chronic medical illness

Healthy Participants (Part A and Part B) and Participants with Primary Sjögren's Syndrome (pSS) (Part C)

- Any major surgery within 4 weeks prior to study drug administration, or any surgery planned during the course of the study

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 137 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 137 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 137 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 137 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 137 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 137 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 137 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 137 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 137 days
  PR interval: The time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QRS interval | Up to 137 days
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QT interval | Up to 137 days
  QT interval: Measured from the beginning of the QRS complex to the end of the T wave
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: QTcF interval | Up to 137 days
  QTcF interval: Corrected QT interval using Fridericia's formula (QTcF)
Incidence of clinically significant changes in physical examination findings | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: C-reactive protein (CRP) | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: Interferon-gamma (IFN-γ) | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: Interleukin-1 beta (IL-1β) | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: Interleukin-6 (IL-6) | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: Interleukin-8 (IL-8) | Up to 137 days
Incidence of clinically significant changes in inflammatory markers: Tumor necrosis factor alpha (TNFα) | Up to 137 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 137 days
Time of maximum observed plasma concentration (Tmax) | Up to 137 days
Area under the plasma concentration-time curve from time zero to time of the last quantifiable concentration (AUC(0-T)) | Up to 137 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Medvin Clinical Research - Metyas, Covina, California, United States
- Local Institution - 0001, Berlin, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome